CLINICAL TRIAL: NCT01652664
Title: A 3 Month, Multicenter, Double-Masked Safety and Efficacy Study of Travoprost Ophthalmic Solution, 0.004% Compared to Timolol (0.5% or 0.25%) in Pediatric Glaucoma Patients
Brief Title: Study of Travoprost Ophthalmic Solution, 0.004% Compared to Timolol (0.5% or 0.25%) in Pediatric Glaucoma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-12-008
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Pediatric Glaucoma; Elevated IOP in Pediatric Patients; Ocular Hypertension in Pediatric Patients
MeSH Terms: conditions — Hydrophthalmos | interventions — Travoprost; Timolol; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost (Experimental): Travoprost 0.004% PQ ophthalmic solution, 1 drop administered in each eye in the evening with travoprost vehicle administered once daily in the morning for 3 months
  Interventions: Drug: Travoprost 0.004% PQ ophthalmic solution; Drug: Travoprost Vehicle
- Timolol (Active Comparator): Timolol, 0.5% or 0.25% ophthalmic solution, 1 drop administered in each eye twice daily (once in the morning and once in the evening) for 3 months
  Interventions: Drug: Timolol, 0.5% or 0.25% ophthalmic solution

INTERVENTIONS:
Drug: Travoprost 0.004% PQ ophthalmic solution
  Arms: Travoprost
Drug: Timolol, 0.5% or 0.25% ophthalmic solution — Patients 2 months to < 3 years of age received 0.25%
  Arms: Timolol
Drug: Travoprost Vehicle — Inactive ingredients used to maintain masking
  Arms: Travoprost

SUMMARY:
The purpose of this study is to evaluate the intraocular pressure (IOP)-lowering efficacy of Travoprost 0.004% POLYQUAD (PQ) ophthalmic solution compared to Timolol ophthalmic solution (0.5% or 0.25%) in pediatric glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pediatric glaucoma or ocular hypertension.
* Qualifying mean IOP at the Eligibility Visit in at least one eye.
* Written informed consent, including assent when applicable, MUST be obtained from the parent or legally authorized representative prior to any procedure specified in the protocol, including screening procedures.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential who are pregnant, intend to become pregnant during the study period, breast feeding, or not using any form of birth control measures.
* History of chronic, recurrent or severe inflammatory eye disease.
* Ocular trauma requiring medical attention within the past 3 months prior to the Screening Visit.
* Ocular infection or ocular inflammation within the past 30 days prior to the Screening Visit.
* Clinically significant or progressive retinal disease.
* Severe ocular pathology (including severe dry eye) that, in the opinion of the Investigator, would preclude the administration of a topical prostaglandin analog or a topical beta-blocker.
* Intraocular surgery in the study eye within 30 days prior to the Screening Visit.
* Any abnormality preventing reliable applanation tonometry.
* Other protocol-defined exclusion criteria may apply.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subha Venkataraman, Clinical Project Lead, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 38 investigational centers in the United States, Germany, Singapore, United Kingdom, Taiwan, Philippines, Spain, Saudi Arabia, Colombia, France, Portugal, Belgium, Poland, Romania, Puerto Rico, and Mexico.
Pre-assignment Details: Of the 184 enrolled, 32 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants (152).
Groups:
- Travoprost: 1 drop administered in each eye in the evening with Travoprost vehicle in the morning for 3 months
- Timolol: 1 drop administered in each eye twice daily (once in the morning and once in the evening) for 3 months; both concentrations of timolol (0.5% and 0.25%, based on age) were combined into a single group.
Period: Overall Study
Arm/Group | Travoprost | Timolol
Started | 77 | 75
Completed | 71 | 74
Not Completed | 6 | 1
Not completed — Treatment Failure | 5 | 1
Not completed — Inadequate IOP control | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants who received study drug and completed at least 1 scheduled on-therapy visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost | Timolol | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Customized [Number; unit: participants]
  2 months to <3 years | 10 | 6 | 16
  3 to <12 years | 40 | 39 | 79
  12 to <18 years | 27 | 30 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 37 | 35 | 72
Intraocular Pressure [Mean (Standard Deviation); unit: mmHg] | 24.7 (4.62) | 24.2 (4.01) | 24.4 (4.32)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in IOP at Month 3
Description: IOP (fluid pressure inside the eye) was assessed using a calibrated tonometer and measured in millimeters of mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye from each participant was chosen as the study eye and only the study eye was used for analysis.
Time Frame: Baseline (Day 0), Month 3
Population: All participants who received study drug and completed at least 1 scheduled on-therapy visit. No imputation was used, therefore the analysis included only observed cases.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Travoprost | Timolol
Number analyzed (Participants) | 71 | 74
mmHg | -5.4 (0.98) | -5.3 (0.93)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (05 Sep 2012 - 25 Mar 2014). This analysis group includes all enrolled participants.
Description: An AE was defined as any untoward medical occurrence in a patient who is administered a study medication, regardless of whether or not the event has a causal relationship with the medication. All AEs were obtained as solicited comments from patients and as observations by the study Investigator as outlined in the study protocol.
Groups:
- Pre-Treatment: All enrolled participants
- Travoprost: All participants who received travoprost with vehicle
- Timolol: All participants who received timolol; both concentrations of timolol (0.5% and 0.25%, based on age) were combined into a single group.
Arm/Group | Pre-Treatment | Travoprost | Timolol
Serious Adverse Events (participants affected / at risk) | 0/184 | 0/77 | 2/75
Other Adverse Events (participants affected / at risk) | 1/184 | 22/77 | 6/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment (N=184) | Travoprost (N=77) | Timolol (N=75)
Keratitis bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment (N=184) | Travoprost (N=77) | Timolol (N=75)
Ocular hyperaemia (Eye disorders) | 0 | 15 | 3
Growth of eyelashes (Eye disorders) | 0 | 5 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 4 | 1
Headache (Nervous system disorders) | 1 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.